CLINICAL TRIAL: NCT04371939
Title: Randomized, Two-arm Single-center Phase II Clinical Trial Comparing the Efficacy and Safety of Romiplostim Versus Eltrombopag in the Treatment of Thrombocytopenia in Patients With Wiskott-Aldrich Syndrome
Brief Title: Efficacy and Safety of Romiplostim Versus Eltrombopag in the Treatment of Thrombocytopenia in Patients With Wiskott-Aldrich Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NCPHOI-2020-03
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Wiskott-Aldrich Syndrome
Keywords: eltrombopag; romiplostim; thrombocytopenia; platelets
MeSH Terms: conditions — Wiskott-Aldrich Syndrome; Thrombocytopenia | interventions — romiplostim; eltrombopag

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I (Romiplostim) (Experimental): Participants will receive romiplostim at an initial dose of 9 µg/kg subcutaneously per week for at least 1 month depending on their response to study drug.
  Patients failing to achieve a complete platelet response cross over to arm II.
  Interventions: Drug: Romiplostim
- II (Eltrombopag) (Experimental): Participants will receive eltrombopag at a dose of 2-3mg/kg daily (ages 0 to 5 years) and 75 mg/daily (>6 years) for at least 1 month depending on their response to study drug.
  Patients failing to achieve a complete platelet response switch to arm I.
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Romiplostim — Participants will receive romiplostim at an initial dose of 9 µg/kg subcutaneously per week for at least 1 month depending on their response to study drug.
  Patients failing to achieve a complete platelet response cross over to arm II.
  Other Names: Nplate
  Arms: I (Romiplostim)
Drug: Eltrombopag — Participants will receive eltrombopag at a dose of 2-3mg/kg daily (ages 0 to 5 years) and 75 mg/daily (>6 years) for at least 1 month depending on their response to study drug.
  Patients failing to achieve a complete platelet response switch to arm I.
  Arms: II (Eltrombopag)

SUMMARY:
This is a prospective, open-label, randomized, two-arm clinical trial conducted to evaluate the safety and efficacy of romiplostim in comparison with eltrombopag in the treatment of thrombocytopenia in patients with Wiskott-Aldrich syndrome

DETAILED DESCRIPTION:
Wiskott-Aldrich syndrome (WAS) is a life-threatening primary immunodeficiency associated with bleeding of variable severity due to severe thrombocytopenia. Considering that the hemorrhagic events are a cause of death in 21% of WAS patients, management of thrombocytopenia constitutes a major challenge. Findings of defective platelet production by megakaryocytes and reduced in vitro pro-platelet formation suggested the possibility of megakaryocyte stimulation by TPO-RAs romiplostim, eltrombopag as a treatment strategy. Each of them has distinct pharmacodynamic, pharmacokinetic properties, different effects on megakaryopoiesis, and might have different efficacy in individual patients.

The aim of this study is to compare the efficacy and safety of romiplostim and another TPO-RA eltrombopag for the treatment of thrombocytopenia in patients with WAS and assess the benefit of switching these molecules in refractory subjects. The patients will be randomized in a 1:1 fashion to receive either romiplostim or eltrombopag.

After enrollment, (see detailed inclusion and exclusion criteria below) subjects under 18 years of age with a confirmed diagnosis of WAS and thrombocytopenia (platelet count of less than 70 x 109/L) will be assigned to receive romiplostim at an initial dose of 9 µg/kg subcutaneously per week or oral eltrombopag at a dose of 2-3mg/kg daily (ages 1 to 5 years) and 75 mg/daily (>6 years) for at least 1 month.

Bleeding severity will be evaluated with a modified World Health Organization (WHO) Bleeding Scale, lab tests (blood counts, biochemical analyses), ECG will be assessed after 30 days of treatment (30 +/- 7 days).

The efficacy of romiplostim/eltrombopag will be defined by the following criteria: complete response -an achievement of the platelet count >100 x 109/L, partial - platelet count at least 30 x 109/L higher than the patient's pretreatment baseline count up to to 100 x 109/L. No response will be defined as not achieving a platelet count of > 30 x 109/L from the baseline count.

Refractory patients will be switched to alternate TPO-RA agonist. Other reasons for switching that are not related to efficacy might include adverse events, active colitis, patient preference.

ELIGIBILITY:
Inclusion Criteria:

* Genetically verified Wiskott-Aldrich syndrome
* Thrombocytopenia (platelet count < 70 x 109/L)
* Age: under 18 years
* Subject/legal representative has signed written informed consent.

Exclusion Criteria:

* Patients, who do not meet the inclusion criteria.
* Any prior history of arterial or venous thrombosis within the past year.
* Arm II (eltrombopag):

  1. abnormal hepatic function -elevated AST/ALT > 1.5 times upper limit of normal within 4 weeks prior to enrollment
  2. Active colitis

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-11-05 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with overall platelet response (complete response + partial response) for romiplostim and eltrombopag group | 1 month (30 day +/- 7 days)
  A complete response will be defined as a platelet count >100 x 109/L, partial - 30 x 109/L higher than the patient's pretreatment baseline count to 100 x 109/L.

SECONDARY OUTCOMES:
Number of participants with bleeding events and severity of bleeding in romiplostim and eltrombopag group | until discontinuation, from at least one month to one year
  The incidence and severity of bleeding events is evaluated with a modified World Health Organization (WHO) Bleeding Scale.
  (G1=Petechiae, epistaxis <30 min, G2=Mild blood loss, hematomas, epistaxis >30 min, melanotic stool G3=Gross blood loss, requiring blood transfusions, G4=Fatal bleeding).
Number of participants with drug related adverse events in each treatment group | until discontinuation, from at least one month to one year
  Adverse events are graded according to Common Terminology Criteria for Adverse Events (CTCAE).
Percentage of patients with overall platelet response (complete response + partial response) after switching from one TPO-RA to another one. | until discontinuation, from at least one month to one year

CONTACTS AND LOCATIONS:
Locations (1):
- Dmitry Rogachev National Research Center of Pediatric Hematology, Oncology and Immunology, Moscow, Russia